CLINICAL TRIAL: NCT04515485
Title: A Volumetric Nomogram for Height, Weight, and Intra Abdominal Volume
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Obstetrics & Gynaecology, Senior Consultant, National University Hospital, Singapore
Other Study IDs: 2019/01152
Record Dates: First submitted 2020-07-01; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Laparoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing laparoscopy: The participants are patients that have undergone the laparoscopic surgery.

SUMMARY:
This is a prospective study to collect a nomogram of intra-abdominal volume correlated with height and weight for O&G patients undergoing minimally invasive surgery.

DETAILED DESCRIPTION:
This is a prospective study from the date of approval of the study for a period of 24 months.

The potential participants are from O&G department who will be undergoing laparoscopy

The participant's height, weight, and total volume of carbon dioxide gas infused into the abdomen are collected from CPSS to create a standard operative pneumoperitoneum of 18mmHg for all patients undergoing laparoscopic procedures.

Patients with an abdomino-pelvic mass, or pelvic masses larger than 12 weeks size, or assessed to have an abdominal mass are excluded. Pregnant and/or breast feeding women are also excluded.

Specific patient identifiers will not be collected into the data collection and are not necessary to the study or to achieving to the objective of the study. Therefore data will not contain any identifiers.

ELIGIBILITY:
Inclusion Criteria:

* O&G patients that are undergoing laparoscopic surgery.

Exclusion Criteria:

* Patients with an abdomino-pelvic mass
* Patients with pelvic masses larger than 12 weeks size
* Patients assessed to have an abdominal mass
* Pregnant and/or breast feeding women

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women going for laparoscopic surgery under the O&G department.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Creation of a nomogram | 2 years
  The study aims to generate a nomogram.
Recording height | 2 years
  in cm
Recording weight | 2 years
  In kg
Recording intra-abdominal volume during surgery | 2 years
  In ml

IPD SHARING:
Plan to Share IPD: No